CLINICAL TRIAL: NCT05623514
Title: Pre-surgical Ultrasound Evaluation for Improving Patient Selection for vNOTES Approach
Brief Title: Ultrasound Evaluation for Improving Patient Selection in vNOTES
Acronym: PUP-VNOTES
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Aya Mohr Sasson, Principle investigator, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HSC-MS-22-0947
Record Dates: First submitted 2022-11-10; First posted 2022-11-21 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Surgery
Keywords: vaginal surgery; trans-vaginal ultrasound examination; sliding sign

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Candidates for vaginal natural orifice trans-luminal surgery approach (Experimental): Candidates for benign gynecological surgery in the vaginal natural orifice trans-luminal surgery approach
  Interventions: Combination Product: Trans-vaginal ultrasound

INTERVENTIONS:
Combination Product: Trans-vaginal ultrasound — Pre-operative trans-vaginal ultrasound in order to evaluate sliding sign between the uterus and the rectum

SUMMARY:
Vaginal Natural Orifice Transluminal Endoscopic Surgery (vNOTES) is an emerging field in minimally invasive surgery. International consensus-based statement was recently published to help guide the basis for adopting vNOTES into clinical practice, including regarding patient selection. It was agreed that women with potential adhesions are not appropriate candidates for vNOTES approach including women with suspected adhesions due to history of severe pelvic inflammatory disease (PID) or endometriosis. However, as some pelvic infections might be asymptomatic, pre-operation imaging might be beneficial to complete improved selection of patients. Moreover, women with previous severe PID or endometriosis might still have favorable pelvic to perform the vNOTES approach. Therefore, we aim to compare pre-operation ultrasound evaluation to operative characteristics and outcomes in women undergoing VNOTES approach surgery.

DETAILED DESCRIPTION:
Vaginal Natural Orifice Transluminal Endoscopic Surgery (vNOTES) is an emerging field in minimally invasive surgery. It has gained the most popularity compared to other transluminal natural orifices such as mouth, rectum or urinary tract. By incorporating the advantages of endoscopic surgery, the vNOTES approach avoids abdominal wall wounds and trocar-related complications. Recent studies report reduced postoperative pain, accelerated postoperative recovery, and decreased postoperative wound infections, as well as achieving highly satisfying cosmetic results. All these made this technique very appealing to surgeons and patients alike.

The feasibility and safety of vNOTES in gynecologic surgeries, was first introduced by Ahn et al. in 2012 that performed vNOTES in ten women with benign uterine adnexal disease. Since then, surgeons have developed the technique in various benign gynecologic surgeries indications. There has been an exponential uptake of the number of surgeons performing vNOTES procedures worldwide with no official guidance to ensure the safe implementation of this technique into gynecological practice. The novelty of the technique is still a matter of concern in sub-populations and different indications.

International consensus-based statement was recently published based on Delphi consensus of expert panel to help guide the basis for adopting vNOTES into clinical practice with respect to eight key domains including patient selection. It was agreed that women with potential adhesions are not appropriate candidates for vNOTES approach including women with a history of a severe PID that is considered contraindication. 97.4% of the experts agreed that it is not necessary to perform a preoperative vaginal culture if the patient is asymptomatic. However, as some pelvic infections might be asymptomatic such as with chlamydia, pre-operation imaging might be beneficial to complete proper patient selection for the vNOTES approach. Moreover, women with previous severe PID infection might still have favorable pelvic to perform the vNOTES approach Aim: To the best of our knowledge no guidelines have been published regarding the pre-operation evaluation and the imaging characteristics. Due to the aforementioned, the aim of our study is to compare pre-operation ultrasound evaluation to operative characteristics and outcomes.

Material and Methods This is a prospective cohort study that will be conducted in a single tertiary medical center. Study population will include all women planned for surgery due to benign indication (adnexectomy/ hysterectomy) that vNOTES approach is considered and have normal vaginal examination (normal mobility of the uterus). Women with history of pelvic radiation, suspected malignancy or combined operations will be excluded from the study.

Intervention:

1. As part of the evaluation at the pre-operation clinics, women will complete vaginal examination to assess for pelvic organs mobility and potential adhesions.
2. Trans-vaginal examination will be completed to evaluate uterus and adnexal characteristics in addition to sliding sign between the uterus to the rectum for the evaluation of the Douglas space.
3. Women with normal ultrasound evaluation and a positive sliding sign will continue with surgery via the vNOTES approach. Women with limited mobility demonstrated on ultrasound will be recommended alternative surgical approaches.

3-Swabs will be collected for potential PID pathogens including chlamydia, gonorrhea, trichomonas and mycoplasma.

4-Operation report- will include information regarding pelvic adhesions, location of the adhesions and abdominal screening (Including diaphragm and liver area). For the study group undergoing vNOTES approach surgery - difficulty to complete anterior or posterior colpotomy will be documented.

Douglas space characteristics of the patients undergoing vNOTES approach surgery will be compared to patients that were ruled from vNOTES approach in order to evaluate the association of the presence or absence of sliding sign on pre operation ultrasound to the clinical findings.

Demographic and clinical characteristics will be collected from women's medical files. Operative and post-operative data will be collected including: operation duration, estimated blood loss, operation complications (hypotension, bladder gut or vascular perforation), post-operative complications (hemorrhage, endometritis, vascular - thromboembolic event, ileus).

ELIGIBILITY:
Inclusion criteria:

- Women planned to undergo surgery for hysterectomy or adnexal indication with normal vaginal examination, that are considered for vNOTES approach.

Exclusion criteria:

* History of radiation to the pelvis
* Malignancy
* Combined current vaginal operation (for the treatment of prolapse/ urinary complaints)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Inclusion criteria include only women undergoing vaginal surgery
Enrollment: 75 (Estimated)
Dates: Start 2022-05-16 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The rate of adhesions/ complicated entry to the Douglas space reported during surgery. | From recruitment in the clinics until one month post operation

SECONDARY OUTCOMES:
Organ damage | From operation until one month post-operation
  Damage caused during the surgery to the bladder, the rectum or blood vessel

CONTACTS AND LOCATIONS:
Overall Officials: Aya Mohr-Sasson, Principal Investigator — The University of Texas Health Science Center, Houston, TX
Locations (1):
- University of Texas, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Jallad K, Walters MD. Natural Orifice Transluminal Endoscopic Surgery (NOTES) in Gynecology. Clin Obstet Gynecol. 2017 Jun;60(2):324-329. doi: 10.1097/GRF.0000000000000280. PMID 28221179
- [Result] Li CB, Hua KQ. Transvaginal natural orifice transluminal endoscopic surgery (vNOTES) in gynecologic surgeries: A systematic review. Asian J Surg. 2020 Jan;43(1):44-51. doi: 10.1016/j.asjsur.2019.07.014. Epub 2019 Aug 20. PMID 31444108
- [Result] Baekelandt J, De Mulder PA, Le Roy I, Mathieu C, Laenen A, Enzlin P, Weyers S, Mol BW, Bosteels JJ. Postoperative outcomes and quality of life following hysterectomy by natural orifice transluminal endoscopic surgery (NOTES) compared to laparoscopy in women with a non-prolapsed uterus and benign gynaecological disease: a systematic review and meta-analysis. Eur J Obstet Gynecol Reprod Biol. 2017 Jan;208:6-15. doi: 10.1016/j.ejogrb.2016.10.044. Epub 2016 Oct 29. PMID 27880893
- [Result] Coomber RS, Sodergren MH, Clark J, Teare J, Yang GZ, Darzi A. Natural orifice translumenal endoscopic surgery applications in clinical practice. World J Gastrointest Endosc. 2012 Mar 16;4(3):65-74. doi: 10.4253/wjge.v4.i3.65. PMID 22442743
- [Result] Ahn KH, Song JY, Kim SH, Lee KW, Kim T. Transvaginal single-port natural orifice transluminal endoscopic surgery for benign uterine adnexal pathologies. J Minim Invasive Gynecol. 2012 Sep-Oct;19(5):631-5. doi: 10.1016/j.jmig.2012.04.001. Epub 2012 Jul 3. PMID 22763314
- [Result] Kapurubandara S, Lowenstein L, Salvay H, Herijgers A, King J, Baekelandt J. Consensus on safe implementation of vaginal natural orifice transluminal endoscopic surgery (vNOTES). Eur J Obstet Gynecol Reprod Biol. 2021 Aug;263:216-222. doi: 10.1016/j.ejogrb.2021.06.019. Epub 2021 Jun 17. PMID 34237485